CLINICAL TRIAL: NCT07262151
Title: The Determination of the Effect of Music on Pain, Anxiety, and Vital Findings in Cancer Patients Treated in Palliative Care Centers : a Quasi-experimental Study
Brief Title: Effect of Music on Pain and Anxiety in Palliative Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Gülsüm Kehribar, Doctor, Karamanoğlu Mehmetbey University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KMU-SHMYO-GK-01
Record Dates: First submitted 2025-11-16; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Cancer Pain; Palliative Care; Anxiety; Music Therapy
Keywords: Anxiety; Cancer; Music; Pain; Palliative care; Vital signs
MeSH Terms: conditions — Neoplasms; Cancer Pain; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: a quasi-experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Intervention Group (Experimental): Before the single-session intervention, the researcher administered the Patient Description Form, STAI, and VAS, and recorded baseline vital signs (Blood Pressure, Pulse Rate, Respiratory Rate, Body Temperature, SpO2).
  The intervention was scheduled between 10:00 a.m. and 5:00 p.m. following the patient's morning analgesic dose. Participants rested comfortably for 30 minutes while listening to music using an MP3 player and headphones. Headphones were used to enhance focus and minimize external noise, with separate devices used for each patient to adhere to infection control standards. Immediately post-intervention (second follow-up), VAS, State Anxiety Inventory, and vital signs were re-measured and recorded.
  Interventions: Other: Music Application
- Control Group (Other): Procedures for the Control Group
  Interventions: Other: Procedures for the Control Group

INTERVENTIONS:
Other: Music Application — Before the single-session intervention, the researcher administered the Patient Description Form, STAI, and VAS, and recorded baseline vital signs (Blood Pressure, Pulse Rate, Respiratory Rate, Body Temperature, SpO2).
  The intervention was scheduled between 10:00 a.m. and 5:00 p.m. following the patient's morning analgesic dose. Participants rested comfortably for 30 minutes while listening to music using an MP3 player and headphones. Headphones were used to enhance focus and minimize external noise, with separate devices used for each patient to adhere to infection control standards. Immediately post-intervention (second follow-up), VAS, State Anxiety Inventory, and vital signs were re-measured and recorded.
  Arms: Music Intervention Group
Other: Procedures for the Control Group — The control group followed the same two-phase data collection protocol as the intervention group (first follow-up). After baseline data collection, the control group was instructed to rest quietly in bed for 30 minutes without any other activity. Immediately after the rest period (second follow-up), the VAS, State Anxiety Inventory, and vital signs were measured and recorded.
  Arms: Control Group

SUMMARY:
Background: Cancer patients receiving palliative care often endure a variety of distressing symptoms, most notably pain and anxiety. Evidence suggests that music offers a symptom-alleviating effect for these patients and can also influence their physiological parameters.

Aim: This investigation was structured as a quasi-experimental study utilizing a pre-test and post-test design with a control group. Its goal was to ascertain the influence of music on pain levels, anxiety states, and vital signs among cancer patients admitted to a palliative care facility.

Methods: Data collection relied on the Patient Demographic Form, the Visual Analog Scale (VAS), the State-Trait Anxiety Inventory (STAI), and a Physiological Parameter Monitoring Form. The intervention group was exposed to relaxing instrumental Turkish music in the maqams of Hicaz and Buselik for a single 30-minute session using MP3 players and headphones, whereas the control group was instructed to observe 30 minutes of bed rest without any other activity. Measurements were taken at baseline (pre-intervention) and immediately after the 30-minute intervention period between 10:00 AM and 5:00 PM following the patient's morning analgesic dose.

DETAILED DESCRIPTION:
Advances in medicine have increased life expectancy, leading to a rise in chronic diseases like cancer, with 14 million new cases annually, projected to reach 22 million by 2030. Cancer patients often face intensive treatments and severe symptoms, including pain and anxiety, highlighting the need for palliative care.

Nurses play a key role in symptom management, using both pharmacological and non-pharmacological methods, including music therapy. Music can stimulate neuroendocrine responses by increasing dopamine and serotonin release, activating the limbic system, increasing endorphin release, and suppressing sympathetic nervous system activity, which contributes significantly to reducing pain and anxiety while also affecting the regulation of vital signs such as blood pressure, pulse, body temperature, respiratory rate, and oxygen saturation.

This study examined the effects of music on pain, anxiety, and vital signs in 32 palliative care cancer patients using a quasi-experimental design with a pretest-posttest control group. The study was conducted between February 2021 and June 2022 at Yozgat City Hospital Palliative Care Center and Karaman Training and Research Hospital Palliative Care Center.

Patients in the intervention group listened to 30 minutes of instrumental Turkish music in the maqams of Hicaz and Buselik; controls rested quietly. The music CD was prepared by experts from the Applied Music Therapy Association (UMTED) and consisted of 13 instrumental works designed to provide relaxation and have a sedative effect. The volume was kept low and the main melody was emphasized.

Data collection took approximately 60 minutes per participant. The intervention was performed between 10:00 AM and 5:00 PM after patients received their first daily analgesic dose. Headphones were used to maintain focus and block extraneous noise, with separate devices for each patient to ensure infection control standards. Further research should explore mechanisms, patient differences, and optimal implementation protocols.

ELIGIBILITY:
Eligibility Criteria:

Inclusion Criteria:

* Diagnosed with cancer
* Receiving palliative care treatment at Yozgat City Hospital or Karaman Training and Research Hospital
* Hospitalized in the palliative care center for at least 7 days
* Aged 18 years or older
* Able to speak and understand Turkish
* Able to communicate verbally
* Oriented to place and time
* No psychiatric disease
* No vision or hearing problems
* Self-reported pain intensity of at least 3 on the Visual Analog Scale in the last 24 hours
* Voluntarily agreed to participate in the study
* Provided written informed consent

Exclusion Criteria:

* Underwent major surgical intervention within the last month
* Currently using another complementary and integrative treatment (e.g., aromatherapy, acupuncture)
* Cognitive impairment preventing questionnaire completion
* Not open to communication
* Died within seven days of hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
• Visual Analog Scale | Baseline (Pre-Intervention) and Immediately Post-Intervention (Total 30-minute intervention period).
  A standard 10 cm tool (Price et al., 1983) where patients mark their current pain level (0 = no pain, 10 = worst possible pain).

SECONDARY OUTCOMES:
State Anxiety (State-Trait Anxiety Inventory - State Subscale) | Baseline (Pre-Intervention) and Immediately After Intervention (30-minute intervention period).
  Developed by Spielberger et al. (1970) and validated for Turkish by Öner and Le Compte (1985). This inventory measures transient (State) anxiety; higher scores indicate higher anxiety. Scores range from 20 to 80. Internal consistency (Cronbach's alpha) in this study was 0.81 for State Anxiety.
Trait Anxiety (State-Trait Anxiety Inventory - Trait Subscale) | Baseline (Pre-Intervention) only.
  Developed by Spielberger et al. (1970) and validated for Turkish by Öner and Le Compte (1985). This inventory measures general (Trait) anxiety; higher scores indicate higher anxiety. Scores range from 20 to 80. Internal consistency (Cronbach's alpha) in this study was 0.76 for Trait Anxiety.

OTHER OUTCOMES:
Systolic Blood Pressure (mmHg) | Baseline (Pre-Intervention) and Immediately Post-Intervention (30-minute intervention period).
  Measured using standardized sphygmomanometer according to clinical standards at baseline and immediately post-intervention.
Diastolic Blood Pressure (mmHg) | Baseline (Pre-Intervention) and Immediately Post-Intervention (30-minute intervention period).
  Measured using standardized sphygmomanometer according to clinical standards at baseline and immediately post-intervention.
Heart Rate (beats per minute) | Baseline (Pre-Intervention) and Immediately Post-Intervention (30-minute intervention period).
  Measured using standardized pulse oximeter at baseline and immediately post-intervention.
Respiratory Rate (breaths per minute) | Baseline (Pre-Intervention) and Immediately Post-Intervention (30-minute intervention period)
  Measured by observation according to clinical standards at baseline and immediately post-intervention.
Body Temperature (degrees Celsius) | Baseline (Pre-Intervention) and Immediately Post-Intervention (30-minute intervention period).
  Measured using a digital thermometer at baseline and immediately post-intervention.
Oxygen Saturation (SpO₂) (%) | Baseline (Pre-Intervention) and Immediately Post-Intervention (30-minute intervention period).
  Measured using standardized pulse oximeter at baseline and immediately post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Tekinsoy Kartın, Principal Investigator — https://sbf.erciyes.edu.tr/
Locations (1):
- Yozgat city hospital, Yozgat, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Witte M, Pinho ADS, Stams GJ, Moonen X, Bos AER, van Hooren S. Music therapy for stress reduction: a systematic review and meta-analysis. Health Psychol Rev. 2022 Mar;16(1):134-159. doi: 10.1080/17437199.2020.1846580. Epub 2020 Nov 27. PMID 33176590

DOCUMENTS (2):
  • Statistical Analysis Plan (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT07262151/SAP_000.pdf
  • Informed Consent Form (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT07262151/ICF_001.pdf